CLINICAL TRIAL: NCT05295394
Title: Dolutegravir-Lamivudine as Dual Therapy in naïve HIV-Infected Patients With Documented M184V Mutation:A Pilot Study
Acronym: PADDLE184V
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment, We did not find participants with the M184V mutation , inclusion criteria , throughout 230 resistance tests carried out
Sponsor: Pedro Cahn (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Pedro Cahn, Scientific director, Fundación Huésped
Organization: Fundación Huésped (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-42
Record Dates: First submitted 2019-10-25; First posted 2022-03-25 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 naive infected patients; dual therapy; M184V mutation
MeSH Terms: interventions — dolutegravir; Lamivudine; Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): dolutegravir 50 mg QD plus lamivudine 300 mg QD
  Interventions: Drug: Dolutegravir plus lamivudine

INTERVENTIONS:
Drug: Dolutegravir plus lamivudine — Dolutegravir 50 mg QD plus lamivudine 300 mg QD
  Other Names: dual therapy

SUMMARY:
The purpose of this study is to evaluate the antiviral efficacy, safety and tolerability of dual therapy with 3TC and DTG as initial therapy among naïve HIV patients with a documented M184V mutation.

DETAILED DESCRIPTION:
This is a pilot study designed to evaluate the antiviral efficacy, safety and tolerability of dual therapy with 3TC and DTG as initial therapy among naïve HIV-1 subjects ≥ 18 years old carrying the M184V mutation

This will be evaluated as the proportion of patients with pVL < 50 copies/mL at week 48 using the ITT-exposed analysis (FDA snaphot).

This study will consist of a screening period of up to 42 days, a 48-week treatment period, followed by a 4-week post-treatment follow-up (FU) period to document late adverse events.

The study will include 20 HIV-1-infected subjects, meeting all inclusion criteria and not meeting any exclusion criteria for this study.

ELIGIBILITY:
Inclusion Criteria

* ≥18 years of age.
* Documented HIV-1 infection defined as a positive rapid test or ELISA plus a plasma HIV-1 RNA ≥5,000 copies/mL or a reactive western blot.
* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB) / Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed (see Appendix 4).
* Naïve to ARV therapies (previous exposure to ARV drugs < 10 days).
* Documented M184V mutation associated with resistance to lamivudine in a previous genotypic test (last 3 months), or at screening.
* HIV RNA at screening visit ≥5,000 copies/mL and <≤100,000 copies/ml
* CD4 ≥200 cells/mL
* Subjects can comply with protocol requirements.
* Subject agrees not to take any medication during the study, including over the counter medicines or herbal preparations, without the approval of the trial physician.
* Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the study.
* The patient is a male or a female who is not breastfeeding or pregnant.
* A female may be eligible to enter and participate in the study if she:

  * is of non-child-bearing potential either defined as post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * is of child-bearing potential with a negative pregnancy test at both screening and day 1, and, agrees to use one of the highly effective methods of contraception to avoid pregnancy described in Appendix 3.

Exclusion Criteria:

Patients will NOT be selected to be part of this study if they meet ANY of the following criteria:

* Alcohol or drug use that might impact on adherence
* Subjects positive for Hepatitis B at screening (+HBsAg), or anticipated need for Hepatitis C virus (HCV) therapy during the study
* Women who are pregnant or breastfeeding, or women who plan to become pregnant in the next 2 years
* interferon, interleukin-2, cytotoxic chemotherapy, Dofetilide (or pilsicainide) or immunosuppressors, antacid drugs containing Ca++ and or Mg++ at study entry
* Grade 4 lab abnormalities
* Primary HIV infection (indeterminate WB or previous negative HIV in the last 6 months
* Opportunistic infection (CDC C category) or other disease and/or clinical condition that, in the investigator's opinion, would compromise the patient's safety or outcome of the study; including malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia
* Subjects who in the investigator's judgment, poses a significant suicidality risk.
* History or presence of allergy to the study drugs or their components or drugs of their class
* Treatment with any of the following agents within 28 days of screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses or treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening or exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product
* Any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound;
* Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN), or ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin)
* Creatinine clearance of <50mL/min via Cockroft-Gault method
* Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
HIV viral load efficacy at week 48 | 48 weeks
  the proportion of patients with pVL < 50 copies/mL at week 48 using the ITT-exposed analysis (FDA snaphot).

SECONDARY OUTCOMES:
HIV viral resistance mutations | At week 48
  the number and the type of HIV resistance mutations among patients that meet the definition of virologic failure .
HIV viral load efficacy at week 24 | week 24 and week 36
  proportion of patients with <400 copies/mL and <50 copies/mL at weeks 24 and 36.
immunological response in CD4 cell count | baseline and week 48
  to measure and compare the absolute values of cd4 cells count in two points, at baseline visit and week 48, in this way we will evaluate the gain or increase of CD4 count cells during the study.
adverse events | baseline to 48 weeks
  To describe frequency, type and severity of clinical and laboratory adverse events based on DAIDS Adverse event grading table , version 2.1
lipid profile change | baseline and week 48
  to measure the change in cholesterol and triglyceride values. we are going to compare the value at the baseline visit and at week 48 for both deteminations, in this way we will evaluate the response or change on the lipid profile.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Fundacion huesped, CABA, Buenos Aires
  - CAICI, Rosario, Santa Fe Province

IPD SHARING:
Plan to Share IPD: Yes
to publish week 48 study results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 month after last patient last visit